CLINICAL TRIAL: NCT02458807
Title: The SENSOR Study: A Mixed-methods Study of SElf-management Checks to Predict exacerbatioNs of Pseudomonas Aeruginosa in Patients With Long-term reSpiratORy Conditions
Acronym: SENSOR
Status: Completed | Type: Observational
Sponsor: Portsmouth Hospitals NHS Trust (Other Government)
Collaborators: University of Portsmouth (Other)
Responsible Party: Sponsor
Other Study IDs: PHT/2014/22
Record Dates: First submitted 2015-05-28; First posted 2015-06-01 (Estimated); Last update posted 2022-09-30 (Actual); Status verified 2022-06

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD); Asthma; Bronchiectasis
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Asthma; Bronchiectasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Daily sputum and urine samples have been collected for study analysis. However we do not plan to extract DNA.
Oversight: Data Monitoring Committee: No

SUMMARY:
The World Health Organisation predicts that lung disease will be the World's third largest killer in the future. This research project is looking to see whether the concept of a "home hospital" using the latest gadgets and iPad technology, can help patients stay well and out of hospital.

Portsmouth Hospitals Trust is collaborating with a Company based in the United Kingdom (UK) who has developed a test to predict when people with lung diseases, such as; asthma, COPD and bronchiectasis, who regularly have chest infections, are about to become poorly with another infection - a form of early warning system. The investigators hope that the test will eventually be able to be used by the patient at home daily, to help self-manage their condition. The test measures whether bacteria are present, in sputum, and in what quantity. This information can be used by the patient's healthcare team to consider providing treatment earlier, thus controlling the infection sooner and reducing the patient's symptoms so that patients can stay at home rather than being regularly admitted to hospital.

Part of this "early warning system" that has been developed by the UK Company includes the daily measurement of a number of indicators of health. These are usually only measured in hospital or by a General Practitioner, but new devices have been made that are simple enough for everyone to use at home.

The investigators will include 30 participants, with non-Cystic Fibrosis (CF) chronic respiratory conditions who will be asked to take daily measurements of their blood pressure, temperature, weight and how well their heart and lungs are working with easy-to-use devices. They will also measure their physically activity with an activity tracker and report their wellness and whether they have taken medication daily. Participants will also be asked to collect a sample of sputum and urine each morning. Taking the samples and measurements should only take between 5-15 minutes each day to carry out.

The sputum and urine will be tested at the hospital and will be recorded and analysed, so that the researchers can learn what happens well before a person with these conditions falls sick and needs hospitalisation.

DETAILED DESCRIPTION:
The purpose of this study is to see whether the concept of a "home hospital" using the latest gadgets and iPad technology, can help patients stay well and out of hospital.

This trial is a single centre, non-randomised, mixed methods study. A longitudinal cohort of patients and their carers (where appropriate) will be asked to collect physiological, biological and disease outcome data over a 6 month period. Both participants and the clinicians responsible for patient care and will have no access to the longitudinal data and this information will not be used to make clinical decisions. The laboratory samples will also be analysed in a blinded manner. These data will then be analysed to develop a model for predicting onset of exacerbations which can be built into a self-monitoring system.

Qualitative methods will be used to explore participant and carer experiences of using the technology and performing daily self-monitoring assessments. The expected duration of participant participation in the cohort will be six months, with an invitation to complete a self-administered questionnaire at baseline to inform a face to face semi-structured interview with patients with, or without carer joint participant at the end of the follow-up period (six months completion).

A total of 30 male and female patients, aged 18 and over will be recruited;

20 patients chronically infected with Pseudomonas Aeruginosa (PA):

• 10 with asthma or COPD and 10 with non-CF bronchiectasis

10 patients with no previously detected PA infection, infected with Haemophilus influenza (HI)

The investigators will also recruit 10 patients plus/minus their carers from the PA group, 5 patients plus/minus their carers from the HI group into the qualitative part of the study.

Methodology:

Potential participants will be recruited from existing asthma, COPD and non-CF bronchiectasis local patient databases in combination with the local laboratory results systems by the clinical care team. Potential participants identified will then be contacted by a member of the local research team who are also the routine clinical care team and invited to attend a specialist research recruitment clinic.

At the research clinic participants will be reviewed by a clinical research fellow and screened for suitability for the study by the research team. Patients and carers will be able to view and try out the self-monitoring devices and tablet-based IT system. Capacity to operate these systems will be assessed as part of the screening. Those who meet eligibility criteria will be given a Participant Information Sheet and/or Carer information sheet if participants wish for their carer to assist them in using the self-monitoring devices and tablet-based IT system daily.

After adequate time to consider and ask questions about the study, participants who are interested in taking part in the trial will be invited to a screening visit where they will be asked to sign a consent form.

At the screening visit, following consent, participants' lung function, blood pressure, oxygen levels, height, weight and BMI will be recorded and general health questions will be asked to gain information on medical history, current medications & smoking status. Participants will also be asked to complete a set of baseline questionnaires.

Following the screening visit (up to 10 days after), the research nurse and an technician from the company ASEPTIKA will deliver and install the study equipment into the participants home and train the participant on how to use all the technology provided. This training visit will take approximately 60 minutes.

Over a period of 6 months, participants will be required to collect a sputum and urine sample daily and store them in the freezer provided, in their own homes. Participants will be trained in sample collection at the screening visit by a member of the research team. The samples will be collected from the participants monthly by the a member of the research team, or participants can bring the samples into hospital at their routine clinic appointments. Participants will also need to measure their weight, blood pressure, oxygen level and lung function and wear an activity monitor daily. These results, as well as a questionnaire, are recorded on the iPad which sends the data via 3G to a central database. The process should take no longer than 15 minutes a day. Participants and clinicians will be blind to the continuous data over the duration of the study but participants will see the values generated daily on the screens of the devices.

During the study participants will attend their normal review with the medical team at 3 and 6 months (study completion) which usually involves lung function, sputum sample for culture and clinical review. These visits will coincide with a short clinic visit to see the research team to complete disease specific and quality of life questionnaires as well as noting any changes to treatment and exacerbations.

Participants and their carers will also have the opportunity to give additional consent to take part in a qualitative interview, at the same time as the main study consent is sought. If consent is attained, participants will be given an extra questionnaire to complete at baseline which will include questions on their expectations and desired outcomes of the study, worries, concerns and any foreseen barriers to compliance. Participants plus or minus their carers may then be selected and invited to take part in 1 semi-structured face-to-face interview, at the end of study (6 months) to discuss what they think about the study and also what they feel and understand about their health. The interviews will either be conducted at the participants' homes or at hospital, depending on their preference and will be conducted by the same research fellow throughout the study to allow consistency. The interviews will take approximately 45-60 minutes depending on what the participant/carer wishes to share. The interview can be terminated at any point the participant/carer wishes to stop and this will not influence their subsequent treatment.

If participants are admitted to hospital during the course of the study they will be asked to take along their iPad and self-monitoring devices with them. If participants forget their iPad a member of the study team will visit the patient on the ward and will assist to collect the patient's daily measurements for the study where appropriate.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female, aged 18 years or above.
* Diagnosed with at least one (or a combination) of the following chronic respiratory conditions: asthma, COPD, non-CF bronchiectasis.
* Previous positive bacterial culture for PA or HI.
* Two or more exacerbations treated with antibiotics with the same pathogen within the last 12 months, one of which must have been within the last 6 months.
* Has been exacerbation free for the previous 4 weeks.
* Producing at least 1ml of sputum daily.
* Must be capable of operating the self-monitoring devices and tablet-based IT system, or have a carer capable of undertaking the measurements and collection, storage and transport of samples.
* Participant is willing and able to give informed consent for participation in the study.

Exclusion Criteria:

* A suspected or confirmed diagnosis of Cystic Fibrosis
* Any condition likely to limit participant survival or adherence during the study period in the judgement of the clinician, for example malignancy, cirrhosis of the liver.
* Currently taking part in any other research study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are self-managing chronic respiratory conditions (apart from CF), and are colonised with either PA or HI and are prone to exacerbation.
Sampling Method: Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2014-08-18; Primary Completion 2015-02-28 (Actual); Study Completion 2015-02-28 (Actual)

PRIMARY OUTCOMES:
Exacerbation | 6 months
  An exacerbation will be defined as the initiation of antimicrobial therapy for respiratory symptoms either at home or on admission, with or without concomitant steroids or admission. For patients who are already on continuous antibiotics, an exacerbation will be defined as starting a course of different antibiotics due to increased symptoms, or an increase or dose or frequency.

SECONDARY OUTCOMES:
Treatment Efficacy | 6 months
  Treatment efficacy will be defined as the day at which antibiotic treatment for that episode is completed.

CONTACTS AND LOCATIONS:
Overall Officials: Prof Anoop Chauhan, Principal Investigator — Portsmouth Hospitals NHS Trust
Locations (1):
- Portsmouth Hospitals NHS Trust, Queen Alexandra Hospital, Portsmouth, Hampshire, United Kingdom

REFERENCES:
- [Background] Pasteur MC, Bilton D, Hill AT; British Thoracic Society Bronchiectasis non-CF Guideline Group. British Thoracic Society guideline for non-CF bronchiectasis. Thorax. 2010 Jul;65 Suppl 1:i1-58. doi: 10.1136/thx.2010.136119. PMID 20627931
- [Background] Murphy TF. The many faces of Pseudomonas aeruginosa in chronic obstructive pulmonary disease. Clin Infect Dis. 2008 Dec 15;47(12):1534-6. doi: 10.1086/593187. No abstract available. PMID 19025364
- [Background] Xie Y, Redmond SJ, Mohktar MS, Shany T, Basilakis J, Hession M, Lovell NH. Prediction of chronic obstructive pulmonary disease exacerbation using physiological time series patterns. Annu Int Conf IEEE Eng Med Biol Soc. 2013;2013:6784-7. doi: 10.1109/EMBC.2013.6611114. PMID 24111301
- See also: NICE Quality Standard for Asthma — http://nice.org.uk/guidance/qs25
- See also: NICE Chronic obstructive pulmonary disease quality standard — http://nice.org.uk/guidance/qs10